CLINICAL TRIAL: NCT06614972
Title: Clinical Outcome of Balloon-Expandable Drug-Eluting Stenting For Patients With Intracranial Atherosclerotic Stenosis: a Prospective, Multicenter, Real-World Registry Study
Brief Title: Balloon-expandable DES for ICAS Registry Study (BDES-ICAS Registry)
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2024-188-B
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Atheroscleroses, Cerebral; Intracranial Atherosclerosis; Ischemia Stroke
Keywords: Intracranial Atherosclerosis Stroke; Drug-eluting stent
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- balloon-expandable drug-eluting stent: Patients were treated with balloon-expandable drug-eluting stent.
  Interventions: Device: Balloon-expandable drug-eluting stent

INTERVENTIONS:
Device: Balloon-expandable drug-eluting stent — Balloon-expandable drug-eluting stent (BDES) is the device comprises of a balloon expandable sirolimus eluting stent and a delivery catheter that features a rapid exchange catheter design with a semi-compliant balloon located at its distal end.

SUMMARY:
To study the clinical outcomes after implantation of balloon-expandable drug-eluting stents in patients with symptomatic intracranial atherosclerotic stenosis in prevention of composite event of any stroke and death within 30 days and ischemic stroke in the territories of the responsible artery from 31 days to 1-year.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, real world, registry study. This study aimed to evaluate the effectiveness of balloon-expandable drug-eluting stents in treating stenosis in the C2-C7 segments of the internal carotid artery and V4 artery which with high prevalence of calcified plaques in ICAD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. According to clinical and angiographic evidence, symptomatic intracranial arteries stenosis within 3 months include vertebral artery V4 segment or internal carotid artery C2-C7 segment, and the degree of diseased arterial stenosis is between 70%~99% (WASID method).
3. Patients have more than 1 episode of symptoms including stroke or transient ischemia attack (TIA) after intensive medical treatment (including antiplatelet therapy, antihypertensive, hypoglycemic and lipid-lowering treatments).
4. Patients have at least 1 risk factor for intracranial atherosclerosis, including previous or existing hypertension, hyperlipidemia, diabetes mellitus, smoking, alcohol consumption, obesity, underlying heart disease, family history of atherosclerotic vascular disease, hyperhomocysteinemia and so on.
5. Baseline mRS score ≤3.
6. Patient or guardian signs informed consent.

Exclusion Criteria:

1. Patients who cannot receive dual antiplatelet therapy due to existing diseases or with server coagulation dysfunction, uncontrolled serious infections, serious systemic diseases, uncontrollable hypertension and other conditions are not suitable for surgery.
2. Patients with aneurysm that cannot be treated in advance or at the same time or are not suitable for surgery.
3. Gastrointestinal disease with active bleeding.
4. Myocardial infarction or massive cerebral infarction within 2 weeks.
5. Patients with known severe allergies or contraindications to heparin, rapamycin, anesthesia and contrast media.
6. Life expectancy <12 months.
7. According to the judgement of the investigator, other situations that are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic intracranial arteries stenosis within 3 months include vertebral artery V4 segment or internal carotid artery C2-C7 segment, and the degree of diseased arterial stenosis is between 70%~99%.
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Any stroke or death within 30 days of implantation or any revascularization procedure OR an ischemic stroke in the territory of the symptomatic intracranial artery between 31 day to 1 year. | 12 months after implantation
  Primary endpoints are composite event of (1) any stroke or death within 30 days after enrollment, (2) any stroke or death within 30 days after revascularization procedure of the qualifying lesion during follow-up, and (3) ischemic stroke in the territory of the qualifying artery from 31 days to 1 year.

SECONDARY OUTCOMES:
Any cerebral events within 1 year | 12 months after implantation
  Cerebral events defined as transient ischemic attack (TIA), ischemic stroke, thrombus and death in the territory of the qualifying artery
Periprocedural events | within 30 days after implantation
  Periprocedural events defined as transient ischemic attack (TIA), ischemic stroke and all-cause death.
In-stent restenosis(ISR) rate | 12 months after implantation
  The ISR is defined as >50% stenosis within or immediately adjacent (within 5 mm) of the implanted stent and >20% absolute luminal loss on angiographic experiment.
Technique success rate | During the procedure
  Technique success was defined as successful arrival of stent to the lesion and subsequent release of the stent delivery system with a residual stenosis of <30%.
Functional outcome measured by modified Rankin Scale and NIH stroke scale (NIHSS) score | Every year after implantation during 5 years
  Modified Rankin Scale (mRS) score and NIHSS score(if need) at every year after implantation during 5 years. The range of modified Rankin Scale was from 0 to 6. 0-No symptoms;1-No significant disability;2-Slight disability;3-Moderate disability;4-Moderately severe disability;5-Severe disability;6 -Dead. A higher score indicates a worse outcome. NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The minimum score is 1 and the maximum score is 20. A higher score indicates a worse outcome.

OTHER OUTCOMES:
In-stent restenosis(ISR) rate | 2-5 years after implantation
  The ISR is defined as >50% stenosis within or immediately adjacent (within 5 mm) of the implanted stent and >20% absolute luminal loss on angiographic experiment.
Any cerebral events | 2-5 years after implantation
  Cerebral events defined as transient ischemic attack (TIA), ischemic stroke, thrombus and death in the territory of the qualifying artery.

CONTACTS AND LOCATIONS:
Overall Officials: Jieqing Wan, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Haven't decided share IPD to other researchers.

REFERENCES:
- [Background] Li G, Wang N, Li X, Ma N, Liu T, Sun Y, Liu P, Miao Z, Zhang Y. Balloon-Mounted versus Self-Expanding Stent Outcomes in Symptomatic Middle Cerebral Artery Stenosis Combined with Poor Collaterals in China: A Multicenter Registry Study. World Neurosurg. 2019 Apr;124:e675-e681. doi: 10.1016/j.wneu.2018.12.189. Epub 2019 Jan 16. PMID 30659967
- [Background] Zhang Y, Rajah GB, Liu P, Sun Y, Liu T, Li X, Miao Z, Li G. Balloon-mounted versus self-expanding stents for symptomatic intracranial vertebrobasilar artery stenosis combined with poor collaterals. Neurol Res. 2019 Aug;41(8):704-713. doi: 10.1080/01616412.2019.1610837. Epub 2019 Apr 28. PMID 31030623
- [Background] Abdollahifard S, Yousefi O, Kamran H, Mowla A. Balloon-mounting stent for intracranial arterial stenosis: A comprehensive and comparative systematic review and meta-analysis. Interv Neuroradiol. 2023 Aug;29(4):466-480. doi: 10.1177/15910199221100620. Epub 2022 May 12. PMID 35549530
- [Background] Bartstra JW, van den Beukel TC, Van Hecke W, Mali WPTM, Spiering W, Koek HL, Hendrikse J, de Jong PA, den Harder AM. Intracranial Arterial Calcification: Prevalence, Risk Factors, and Consequences: JACC Review Topic of the Week. J Am Coll Cardiol. 2020 Sep 29;76(13):1595-1604. doi: 10.1016/j.jacc.2020.07.056. PMID 32972537
- [Background] Ma N, Zhang Y, Shuai J, Jiang C, Zhu Q, Chen K, Liu L, Li B, Shi X, Gao L, Liu Y, Wang F, Li Y, Liu T, Zheng H, Mo D, Gao F, Wang Y, Wang Y, Feng L, Miao Z. Stenting for symptomatic intracranial arterial stenosis in China: 1-year outcome of a multicentre registry study. Stroke Vasc Neurol. 2018 May 7;3(3):176-184. doi: 10.1136/svn-2017-000137. eCollection 2018 Sep. PMID 30294474